CLINICAL TRIAL: NCT02104921
Title: Innovative Ultrasound Technology in Neuromuscular Disease
Acronym: AQUIRe
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Seward Rutkove, Professor of Neurology, Beth Israel Deaconess Medical Center
Other Study IDs: 2012P000364; 2K24NS060951 (NIH)
Record Dates: First submitted 2014-03-31; First posted 2014-04-07 (Estimated); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Amyotrophic Lateral Sclerosis; Muscular Dystrophy; Radiculopathy; Myopathy; Polyneuropathy and Mononeuropathies; Trauma Injury; Orthopedic Disorder
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Muscular Dystrophies; Radiculopathy; Muscular Diseases; Polyneuropathies; Mononeuropathies; Accidental Injuries; Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Neuromuscular Disease Patients: Amyotrophic lateral sclerosis patients, myopathy patients, muscular dystrophy patients, myasthenia gravis patients, radiculopathy patients, mononeuropathy patients
- Healthy volunteers

SUMMARY:
This study is utilizing ultrasound measurement to measure neuromuscular disease status in adult patients. The hypothesis is the by quantifying ultrasound data, it is possible that ultrasound can be utilized as a tool to determine if a disease is responding to therapy or progressing.

ELIGIBILITY:
Inclusion Criteria:

* History of a well-defined, localized or generalized neuromuscular condition producing weakness or muscle atrophy, including disuse atrophy.

Exclusion Criteria:

* Multiple generalized neuromuscular conditions.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with any neuromuscular disorder (i.e. primary nerve or muscle disease), both localized and generalized, producing some degree of weakness or disability.
Sampling Method: Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2013-12-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Quantitative ultrasound data, including quantified grayscale data and backscattered acoustic data | 1 year
  Ultrasound data will be collected on multiple muscles in each person. The images will then be quantified using either 1. A grayscale technique in which the images themselves are analyzed via standard image software (e.g., Adobe Photoshop) as to level of echo intensity in a pre-specific region of interest or 2. the raw quantified backscatter data is captured by the transducer, expressed as a unit of power, in the same pre-specified area of interest

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States